CLINICAL TRIAL: NCT03419780
Title: Can a Single-unit Blood Transfusion Protocol in Obstetrics Reduce Total Number of Units Transfused? A Randomized, Controlled Trial
Brief Title: SMaRT Blood: Single-unit Versus Multiple-unit Packed Red Blood Cell Transfusion in Non-acute Postpartum Anemia
Acronym: SMaRTBlood
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 829141
Record Dates: First submitted 2018-01-17; First posted 2018-02-05 (Actual); Results first posted 2020-11-04 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Postpartum Anemia Nos
MeSH Terms: interventions — Blood Transfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Single-Unit Blood Transfusion Protocol (Active Comparator): In this arm, patients receive a 1 unit pRBC transfusion with the plan for post-transfusion blood count at 4-6 hours post-transfusion and clinical reassessment.
  Interventions: Biological: Blood Transfusion
- Multiple-Unit Blood Transfusion Protocol (Active Comparator): In this arm, patients receive 2 units of pRBCs, followed by 4-6 hour post-transfusion blood count and clinical reassessment.
  Interventions: Biological: Blood Transfusion

INTERVENTIONS:
Biological: Blood Transfusion — Patients are randomized to receive 1 or 2 units of packed red blood cells for initial transfusion.

SUMMARY:
There is a paucity of data on management of non-acute postpartum anemia. Although blood transfusions were historically initiated with 2 units, the most recent recommendation from the American Association of Blood Banks is to begin with 1 unit. As no randomized controlled trials have been performed in obstetrics, the investigators propose a randomized, controlled trial in non-acute postpartum anemia comparing single- versus multiple-unit transfusion by total numbers of units transfused and maternal morbidity.

DETAILED DESCRIPTION:
Postpartum hemorrhage (PPH), which accounts for 30% of all direct maternal deaths, is the single most important cause of maternal morbidity and mortality across the globe and is a focus of attention of national organizations such as the Council for Patient Safety in Women's Health in recent years. Yet, there remains a paucity of data on the appropriate management of non-acute postpartum anemia.

It is common practice in obstetrics to offer a transfusion of packed red blood cells (pRBCs) to women with a hemoglobin (Hb) value less than 7 g/dL (hematocrit less than 20%) and to symptomatic women with even higher hemoglobin levels. Although transfusions were historically initiated with 2 units of pRBCs, the most recent recommendation from the American Association of Blood Banks (AABB) for a stable patient is to begin with 1 unit and reassess. However, while surgical data has successfully demonstrated that liberal blood transfusion increases morbidity and mortality in comparison to restricted transfusion, no randomized controlled trials have been performed in obstetrics to demonstrate superiority of a single-unit transfusion protocol.

The investigators propose a randomized, controlled trial in non-acute postpartum anemia comparing single-unit versus multiple-unit transfusion by total numbers of units transfused and maternal morbidity at the University of Pennsylvania with the hypothesis that single-unit transfusions can reduce the number of units transfused without increasing maternal morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Women over 18
* Willing and stable to give consent
* > 6 hours postpartum from any mode of delivery
* Determined by their physician to require blood transfusion either by:

  * Hb <7g/dL OR
  * >7g/dL with any sign or symptom of anemia such as fatigue, dizziness, tachycardia, or hypotension
* Agreed to accept blood transfusion
* No contraindications to blood transfusion

Exclusion Criteria:

* hemoglobinopathies
* patients with an ejection fraction <35%
* Hb <5 g/dL
* HR > 130 bpm, BP < 80/40

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Eligibility is determined by delivery of a fetus.
Enrollment: 66 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sindhu K Srinivas, MD MSCE, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Carson JL, Stanworth SJ, Dennis JA, Trivella M, Roubinian N, Fergusson DA, Triulzi D, Doree C, Hebert PC. Transfusion thresholds for guiding red blood cell transfusion. Cochrane Database Syst Rev. 2021 Dec 21;12(12):CD002042. doi: 10.1002/14651858.CD002042.pub5. PMID 34932836
- [Derived] Hamm RF, Perelman S, Wang EY, Levine LD, Srinivas SK. Single-unit vs multiple-unit transfusion in hemodynamically stable postpartum anemia: a pragmatic randomized controlled trial. Am J Obstet Gynecol. 2021 Jan;224(1):84.e1-84.e7. doi: 10.1016/j.ajog.2020.07.007. Epub 2020 Jul 9. PMID 32652065

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single-Unit Blood Transfusion Protocol | Multiple-Unit Blood Transfusion Protocol
Started | 33 | 33
Completed | 33 | 33
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Single-Unit Blood Transfusion Protocol | Multiple-Unit Blood Transfusion Protocol | Total
Number analyzed (Participants) | 33 | 33 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 29 (6) | 29 (6) | 29 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 33 | 66
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 32 | 32 | 64
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 26 | 24 | 50
  White | 4 | 7 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Hemoglobin level at randomization [Mean (Standard Deviation); unit: g/dL] | 6.8 (0.6) | 7.0 (0.6) | 6.9 (0.6)

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Units Transfused
Description: To determine if there is a difference between single-unit and multiple-unit transfusion protocols in total number of units transfused
Time Frame: From randomization until discharge from admission for delivery, an average of 2-3 days
Measure: Mean (Standard Deviation); unit: units of blood
Arm/Group | Single-Unit Blood Transfusion Protocol | Multiple-Unit Blood Transfusion Protocol
Number analyzed (Participants) | 33 | 33
units of blood | 1.2 (0.5) | 2.1 (0.4)
Statistical Analysis 1: Comparison: Single-Unit Blood Transfusion Protocol vs Multiple-Unit Blood Transfusion Protocol; Test type: Superiority; p < 0.001, t-test, 2 sided

2. Secondary Outcome: Length of Stay
Description: To determine if there is a difference between single-unit and multiple-unit transfusion protocols in length of stay in days
Time Frame: From randomization until discharge from admission for delivery, an average of 2-3 days
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Single-Unit Blood Transfusion Protocol | Multiple-Unit Blood Transfusion Protocol
Number analyzed (Participants) | 33 | 33
Days | 3.1 [2.5 to 3.8] | 3.4 [2.4 to 4.1]
Statistical Analysis 1: Comparison: Single-Unit Blood Transfusion Protocol vs Multiple-Unit Blood Transfusion Protocol; Test type: Superiority; p = 0.79, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Number of Participants Exclusively Breastfeeding at 4-9 Weeks Postpartum
Description: To determine if there is a difference between single-unit and multiple-unit transfusion protocols in exclusive breastfeeding rates at 4-9 weeks postpartum.
Time Frame: At 4-9 weeks after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Single-Unit Blood Transfusion Protocol | Multiple-Unit Blood Transfusion Protocol
Number analyzed (Participants) | 29 | 27
Participants | 16 | 15
Statistical Analysis 1: Comparison: Single-Unit Blood Transfusion Protocol vs Multiple-Unit Blood Transfusion Protocol; Test type: Superiority; p = 0.89, Chi-squared

4. Secondary Outcome: Rate of Depression
Description: • To determine if there is a difference between single-unit and multiple-unit transfusion protocols in Edinburgh Postnatal Depression Scale score at 4-9 weeks postpartum. EPDS scores range from 0-30, with higher scores (particularly above 10) are indicative of depression.
Time Frame: 4-9 weeks after randomization
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Single-Unit Blood Transfusion Protocol | Multiple-Unit Blood Transfusion Protocol
Number analyzed (Participants) | 33 | 33
score on a scale | 4 [1 to 11] | 5.5 [2 to 8]
Statistical Analysis 1: Comparison: Single-Unit Blood Transfusion Protocol vs Multiple-Unit Blood Transfusion Protocol; Test type: Superiority; p = 0.34, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Rate of Fatigue
Description: • To determine if there is a difference between single-unit and multiple-unit transfusion protocols in Multidimensional Fatigue Inventory scores at 4-9 weeks postpartum. This score ranges from 0-140 with higher scores indicating worse fatigue.
Time Frame: 4-9 weeks after randomization
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Single-Unit Blood Transfusion Protocol | Multiple-Unit Blood Transfusion Protocol
Number analyzed (Participants) | 33 | 33
score on a scale | 44 [34 to 55] | 53 [38 to 70]
Statistical Analysis 1: Comparison: Single-Unit Blood Transfusion Protocol vs Multiple-Unit Blood Transfusion Protocol; Test type: Superiority; p = 0.13, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Maternal Attachment Inventory Scores
Description: • To determine if there is a difference between single-unit and multiple-unit transfusion protocols in Maternal Attachment Inventory scores at 4-9 weeks postpartum. The possible range of scores is 26-104. Higher scores indicate higher maternal attachment to the infant.
Time Frame: 4-9 weeks after randomization
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Single-Unit Blood Transfusion Protocol | Multiple-Unit Blood Transfusion Protocol
Number analyzed (Participants) | 33 | 33
score on a scale | 104 [102 to 104] | 104 [102 to 104]
Statistical Analysis 1: Comparison: Single-Unit Blood Transfusion Protocol vs Multiple-Unit Blood Transfusion Protocol; Test type: Superiority; p = 0.55, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Infection Rate
Description: Development of any deep or superficial infection
Time Frame: From randomization until 4-9 week postpartum visit
Measure: Number; unit: participants
Arm/Group | Single-Unit Blood Transfusion Protocol | Multiple-Unit Blood Transfusion Protocol
Number analyzed (Participants) | 33 | 33
participants | 2 | 1
Statistical Analysis 1: Comparison: Single-Unit Blood Transfusion Protocol vs Multiple-Unit Blood Transfusion Protocol; Test type: Superiority; p = 1.00, Chi-squared

ADVERSE EVENTS:
Time Frame: Randomization until the time of the postpartum visit which occurred between 4 and 9 weeks after delivery.
Description: The need for additional blood products and prolonged length of stay will not be considered adverse events as they represent possible issues related to the single-unit blood transfusion protocol. Adverse Events will be obtained by review of the subject's electronic medical record.
Arm/Group | Single-Unit Blood Transfusion Protocol | Multiple-Unit Blood Transfusion Protocol
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/33
Other Adverse Events (participants affected / at risk) | 0/33 | 1/33
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single-Unit Blood Transfusion Protocol (N=33) | Multiple-Unit Blood Transfusion Protocol (N=33)
Unrelated transfer to the ICU (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2019-01-15): https://cdn.clinicaltrials.gov/large-docs/80/NCT03419780/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2018-02-15): https://cdn.clinicaltrials.gov/large-docs/80/NCT03419780/Prot_SAP_001.pdf